CLINICAL TRIAL: NCT06277141
Title: The Vitality Mammography Study - Testing the Effectiveness of a Booking Platform on Receipt of Screening Mammography - a Randomized Controlled Trial.
Brief Title: The Vitality Mammography Messaging Study
Acronym: VMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wits Health Consortium (Pty) Ltd (Other)
Collaborators: Discovery Vitality (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: M230742
Record Dates: First submitted 2023-10-27; First posted 2024-02-26 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer Female
Keywords: Mammography; Screening; Social Media

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Standard message (Experimental): standard message reminder to screen for breast cancer.
  Interventions: Behavioral: Standard message
- Radiology Booking Site Link (Experimental): Message with an online link to a radiology practice booking site.
  Interventions: Behavioral: Radiology booking site link.
- Radiology practice telephone numbers (Experimental): Message with a list and telephone numbers of radiology practices.
  Interventions: Behavioral: Radiology practice telephone numbers
- Control - no message (No Intervention): Participants will not receive any messaging regarding mammography.
- Radiology booking site link and telephone numbers. (Experimental): Message with a direct online link to a radiology practice booking site and telephone numbers of radiology practices.
  Interventions: Behavioral: Radiology site link and telephone numbers

INTERVENTIONS:
Behavioral: Standard message — Participants will receive standard messaging based on the Cancer Association of South Africa (CANSA) recommendation on breast cancer screening and a reminder to screen for breast cancer.
  Arms: Standard message
Behavioral: Radiology booking site link. — Participants will receive a reminder to screen for breast cancer with a direct online link to a radiology practice booking site.
  Arms: Radiology Booking Site Link
Behavioral: Radiology practice telephone numbers — Participants will receive a reminder to screen for breast cancer together with a list and telephone numbers of radiology practices
  Arms: Radiology practice telephone numbers
Behavioral: Radiology site link and telephone numbers — Participants will receive a reminder to screen for breast cancer with a direct online link to a radiology practice booking site and a list and telephone numbers of radiology practices
  Arms: Radiology booking site link and telephone numbers.

SUMMARY:
The investigators will be conducting a randomized controlled trial amongst members of a Wellness Program to test receipt of mammogram using the Whatsapp social media platform and testing various messages.

DETAILED DESCRIPTION:
The investigators will be conducting a randomised control trial to test the efficacy of WhatsApp messages to increase receipt of mammography amongst eligible women who are members of the Vitality health promotion programme and are also on the Discovery Health Medical Scheme. The study will test a message that 1) has a link to a platform created by the Radiology Society of South Africa which allow members to select a range of practices to book a mammogram, against 2) a message that gives names and telephone numbers of Radiology practices in a 5 km radius of the members home address, against 3) a group with a link to an online platform as well as telephone numbers of radiology practices, against 4) a group where a standard message reminding to go for mammogram will be sent, but without names and telephone numbers of the radiology practices, against 5) a control group where no messages relating to mammography will be sent.

ELIGIBILITY:
Inclusion Criteria:

* Females aged 50 to 75 years, who are members of the Discovery Health Medical Plan and who are also members of Vitality and who have not had a screening mammogram in the preceding three years and who have not previously been diagnosed with breast cancer.

Exclusion Criteria:

* CPA Blocks
* If member's address location, based on their Discovery profile, was further than 5km radius to the Radiologist practice

Ages: 50 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7655 (Actual)
Dates: Start 2023-09-27 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Comparison of mammography screening rates using WhatsApp | Five months
  Comparison of mammography screening rates using an online radiology booking platform, a message with a radiology practice number, to a standard message, all delivered by WhatsApp.

CONTACTS AND LOCATIONS:
Overall Officials: Adele Walker, Principal Investigator — Discovery
Locations (1):
- University of Witwatersrand, Johannesburg, Gauteng, South Africa

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data will be shared with Wits collaborators
Supporting Information: Study Protocol, SAP, CSR
Time Frame: February 2024 and data will be available until February 2025
Access Criteria: Only select individuals will have access to the data. Data will be password protected.